CLINICAL TRIAL: NCT05232695
Title: Comparison of Brown Fat Tissue-related Hormone Levels in Metabolically Healthy and Unhealthy Obese Individuals
Brief Title: Brown Fat Tissue Related Hormone Levels in Metabolically Healthy and Unhealthy Obese Individuals
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Hacer Hicran Mutlu, Assoc. Prof., Istanbul Medeniyet University
Other Study IDs: Batokines-09
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Metabolically Healthy Obesity
Keywords: metabolically healthy obese; irisin; FGF21; NRG4
MeSH Terms: conditions — Obesity, Metabolically Benign

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples to assess irisin, FGF-21 and NRG4 concentrations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metabolically healthy obese individuals: Individuals who have a body mass index equal or higher than 30 kg/m2, no medication usage, who have only high waist circumference without any other metabolic syndrome criteria.
  Interventions: Diagnostic Test: metabolically healthy obese
- metabolically unhealthy obese individuals: Individuals who have a body mass index equal or higher than 30 kg/m2, no medication usage, who have more than one metabolic syndrome criteria (as defined below) including high waist circumference.
  Interventions: Diagnostic Test: metabolically healthy obese

INTERVENTIONS:
Diagnostic Test: metabolically healthy obese — Obese individuals will be divided into 2 groups as metabolic healthy and unhealthy obese, and their batokine concentrations will be compared.
  Other Names: metabolically unhealthy obese

SUMMARY:
There are two types of adipose tissue in humans, white and brown adipose tissue. While the main task of white adipose tissue is energy storage, the main task of brown adipose tissue is energy expenditure. It was previously thought that only infants have brown adipose tissue, however today it is known that metabolically active brown adipose tissue exists in adult humans as well. Brown adipose tissue contributes to metabolic health through both energy expenditure and the cytokines they secrete.

Although obesity is frequently associated with many metabolic dysfunctions and cardiometabolic diseases such as insulin resistance, prediabetes, atherogenic dyslipidemia, metabolic syndrome, some obese individuals have been defined as metabolically healthy obese. The mechanisms underlying the formation of the metabolic healthy obese phenotype are not well understood. In experimental animal studies, it has been suggested that the molecular phenotype of adipose tissue is an important factor affecting metabolic health in obese individuals. One of the most important factors affecting the molecular phenotype of adipose tissue is the browning potential of adipose tissue. Based on this hypothesis, in this study it is aimed to investigate whether the browning of white adipose tissue has an effect on determining the metabolic phenotype of metabolically healthy and unhealthy obese individuals with the same amount of adipose tissue.

It is known that irisin, FGF21 and NRG4 are hormones that have the ability to brown the white adipose tissue. In our study, it was aimed to investigate whether there is a difference in serum FGF21, irisin and Neuregulin4 (NRG4) levels, which have brown adipose tissue browning potential, in metabolically healthy and unhealthy obese. In this way, it will be found out whether serum FGF21, irisin and NRG4 hormones, which have a browning effect on white adipose tissue, have an effect on the metabolic health of obese individuals and whether these hormones can be a treatment target.

In this project, participants who have BMI ≥30 kg/m2 and no criteria other than metabolic syndrome criteria, except increased waist circumference (blood pressure ≥130/85 mmHg, fasting blood glucose ≥100 mg/dl, triglyceride ≥150 mg/dl, HDL <40mg/dl in men, <50 mg/dl in women) and those without prediabetes will be defined as metabolically healthy obese, on the other hand other obese individuals will be defined as metabolic unhealthy. 10 ml blood samples will be taken from at least 60 metabolically healthy and 60 metabolically unhealthy participants. Serum FGF21, irisin and NRG4 levels will be measured and their levels in metabolically healthy and unhealthy obese individuals will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥30
* Body fat percentage ≥30% in women, ≥25% in men

Exclusion Criteria:

* antidiabetic medication usage
* antihypetrensive mediaction usage
* lipid lowering medication usage
* pregancy
* hypo/hyperthyroidism
* steroid usage
* benign/ malign tumor diagnosis
* liver disease
* secondary causes of obesity

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: individuals who attend to the hospital's obesity outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Specific batokine concentrations in metabolically healthy end unhealthy obese individuals. | 1 year
  The participants' irisin, FGF-21 and NRG-4 levels will be measured to compare their concentrations in metabolically healthy and unhealthy obese individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Mutlu, Assoc. Prof., Principal Investigator — Istanbul Medeniyet University Goztepe Prof Dr Suleyman Yalcın City Hospital
Locations (1):
- Istanbul Medeniyet University Goztepe Prof Dr Suleyman Yalcın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided

REFERENCES:
- [Background] White JD, Dewal RS, Stanford KI. The beneficial effects of brown adipose tissue transplantation. Mol Aspects Med. 2019 Aug;68:74-81. doi: 10.1016/j.mam.2019.06.004. Epub 2019 Jun 21. PMID 31228478